CLINICAL TRIAL: NCT01793142
Title: Post Marketing Surveillance For General Drug Use To Assess The Safety And Efficacy Profile Of Viviant In Usual Practice.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1781047
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; postmenopausal; SERM
MeSH Terms: conditions — Osteoporosis | interventions — bazedoxifene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Viviant treatment group: Viviant treatment group
  Interventions: Drug: Viviant

INTERVENTIONS:
Drug: Viviant — Viviant (Bazedoxifene) 20mg once daily

SUMMARY:
This survey is conducted for preparing application material for re examination under the Pharmaceutical Affairs Laws and its Enforcement Regulation, and assessing the safety and efficacy profiles of VIVIANT in usual practice according to the Re-examination Regulation for New Drugs

DETAILED DESCRIPTION:
continuous enrollment

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal osteoporosis and osteopenia patients

Exclusion Criteria:

* Patients with active or past history of venous thromboembolic events including deep vein thrombosis,
* Patients with pulmonary embolism and retinal vein thrombosis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Postmenopausal osteoporosis and osteopenia patients
Sampling Method: Non-Probability Sample
Enrollment: 3430 (Actual)
Dates: Start 2013-10-24 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- South Korea (60):
  - Inje University Haeundae Paik Hospital, Haeundae-gu, Busan
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul, Capital Metropolitan
  - Dankook University Hospital, Cheonan-si, Chuncheongnam-do
  - Yonsei University Wonju College of Medicine, Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Sejong Hospital, Bucheon-si, Gyeonggi-do
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Inje University Ilsanpaik Hospital, Goyang-si, Gyeonggi-do
  - National Health Insurance Corporation Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Il-San Gaspel Hospital, Goyang-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Wonkwang University Sanbon Hospital, Gunpo, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - St. Vincent's Hospital-The Catholic University of Korea, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Dongguk University Gyeongju Hospital, Gyeongju, Gyeongsangbuk-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Yangsan Hospital-Pusan National University, Yangsan, Gyeongsangnam-do
  - Wonkwang University Hospital, Iksan-si, Jeollabuk-do
  - Soon Chun Hyang University Hospital Seoul, Seoul, Korea
  - Eulji University Hospital, Daejeon, Republic of Korea
  - Severance Hospital, Yonsei University Health System, Seoul, Seodaemun-gu
  - Hanyang University Medical Center, Seongdong-ku, Seoul
  - Sung Mo O.S, Taebang-dong, Seoul
  - Pusan National University Hospital, Busan
  - Dongrae Bongseng Hospital, Busan
  - Centum Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National Univ. Hospital, Daegu
  - Daejeon St. Mary's Hospital-The Catholic University of Korea, Daejeon
  - Chungnam National University Hospital (CNUH), Daejeon
  - Wonju Severance Christian Hospital, Gangwon-do
  - Hosan OS Clinic, Goyang-si
  - Gwangju Veterans Hosptial, Gwangju
  - Donguk University Gyeongju Hospital, Gyoungju
  - Gachon University Gil Hospital, Incheon
  - Christian Internal Medicine Clinic, Incheon
  - Inje University Sanggye Paik Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yeonsei University Health System, Seoul
  - Severance Hospital-Yonsei University College of Medicine, Seoul
  - Cheil General Hospital & Women's Healthcare Center, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center-University of Ulsan College of Medicine, Seoul
  - Asan Medical Center, Seoul
  - Seoul St. Mary Hospital, The Catholic University of Korea, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Choongmu Hospital, Seoul
  - Seoul Medical Center, Seoul
  - Kwangmyeong Sungae Hospital, Seoul
  - Hongik Hospital, Seoul
  - Jung Dong Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Viviant Tablet 20 mg: Participants who received Viviant tablet 20 milligram (mg) once daily orally as a part of routine clinical practice for the first time, were observed for up to a maximum of 6 months. The dose and frequency of Viviant tablet was according to the treating physician as per the approved product labelling.
Period: Overall Study
Arm/Group | Viviant Tablet 20 mg
Started | 3430
Treated | 3423
Completed | 3423
Not Completed | 7
Not completed — Randomized not treated | 7

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received Viviant 20 mg tablet at least once and completed the follow up.
Arm/Group | Viviant Tablet 20 mg
Number analyzed (Participants) | 3423
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean Age | 69.51 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3423
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight Continuous [Mean (Standard Deviation); unit: kilograms] | 55.12 (8.26)
Height Continuous [Mean (Standard Deviation); unit: centimeter] | 153.56 (5.87)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose of Viviant 20 mg tablet, that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline, up to 28 days after last dose of Viviant 20 mg (up to 6 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Viviant Tablet 20 mg
Number analyzed (Participants) | 3423
Participants
  AEs | 209
  SAEs | 17

2. Secondary Outcome: Overall Efficacy Evaluation of Viviant 20 mg Tablet
Description: Efficacy evaluation of Viviant 20 mg tablet was carried out on the basis of the assessment of clinical response by the treating physician. Clinical response among participants were assessed by the physician as improved, no change, worsened and unevaluable for efficacy.
Time Frame: Baseline up to 3 months
Population: Efficacy analysis set included all participants who received Viviant 20 mg tablet at least once and completed evaluation of efficacy endpoints at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Viviant Tablet 20 mg
Number analyzed (Participants) | 3111
Participants
  Improved | 1283
  No change | 1814
  Worsened | 14
  Unevaluable | 0

3. Secondary Outcome: Number of Participants With Osteoporosis Related Fractures
Time Frame: Baseline up to 3 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Viviant Tablet 20 mg
Number analyzed (Participants) | 3111
Participants | 4

4. Secondary Outcome: Number of Participants With Abnormal Dual Energy X-Ray Absorptiometry (DXA)
Description: DXA is established standard for measuring bone mineral density. Criteria for abnormality was based on investigator's discretion.
Time Frame: Baseline up to 3 months
Population: Efficacy analysis set included all participants who received Viviant 20 mg tablet at least once and completed evaluation of efficacy endpoints at least once. Here, "N (number of participants analyzed)" signifies number of participants analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Viviant Tablet 20 mg
Number analyzed (Participants) | 62
Participants | 7

5. Primary Outcome: Number of Participants With Treatment Related Adverse Drug Reactions (ADRs), Serious ADRs, and Unexpected ADRs
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both serious and non-serious AEs. All AEs, except for those with causal relationship to the study drug assessed as "unlikely" or "no", were considered as ADRs. Unexpected AEs/ADRs were classified by medical review with reference to the local product document and confirmed by Pfizer. Treatment related ADRs included all ADRs with causality related to treatment as judged by the investigator.
Time Frame: Baseline up to 28 days after last dose of Viviant 20 mg (up to 6 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Viviant Tablet 20 mg
Number analyzed (Participants) | 3423
Participants
  ADRs | 132
  Serious ADRs | 3
  Unexpected ADRs | 93

6. Secondary Outcome: Number of Participants With Abnormal X-ray Result
Description: Criteria for abnormality was based on investigator's discretion.
Time Frame: Baseline up to 3 months
Population: Efficacy analysis set included all participants who received Viviant 20 mg tablet at least once and completed evaluation of efficacy endpoints at least once. Here, "N" signifies number of participants analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Viviant Tablet 20 mg
Number analyzed (Participants) | 40
Participants | 0

7. Secondary Outcome: Number of Participants With Abnormal Bone Mineral Density Result
Description: A bone mineral density test examines segments of bone through X-rays to detect osteoporosis. Criteria for abnormality was based on investigator's discretion.
Time Frame: Baseline up to 3 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Viviant Tablet 20 mg
Number analyzed (Participants) | 1
Participants | 0

8. Secondary Outcome: Number of Participants With Abnormal Biochemical Markers of Bone Turnover
Description: In this study biochemical markers of bone turnover included C-telopeptide of collagen cross links (CTX), osteocalcin and bone specific alkaline phosphatase. Criteria for abnormality was based on investigator's discretion.
Time Frame: Baseline up to 3 months
Population: Efficacy analysis set included all participants who received Viviant 20 mg tablet at least once and completed evaluation of efficacy endpoints at least once. Here, "n (number analyzed)" signifies the number of participants with available data for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | Viviant Tablet 20 mg
Number analyzed (Participants) | 3111
Participants
  CTX: number analyzed (Participants) | 125
  CTX | 0
  Osteocalcin: number analyzed (Participants) | 20
  Osteocalcin | 0
  Bone specific alkaline phosphatase: number analyzed (Participants) | 1
  Bone specific alkaline phosphatase | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of Viviant 20 mg tablet (up to 6 months)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Viviant Tablet 20 mg
All-Cause Mortality (participants affected / at risk) | 1/3423
Serious Adverse Events (participants affected / at risk) | 17/3423
Other Adverse Events (participants affected / at risk) | 192/3423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Viviant Tablet 20 mg (N=3423)
SPINAL STENOSIS (Nervous system disorders) | 1
BRADYCARDIA (Cardiac disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
DEATH (General disorders) | 1
FATIGUE (General disorders) | 1
FEVER (General disorders) | 1
OEDEMA GENERALISED (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
PYELONEPHRITIS (Infections and infestations) | 3
FRACTURE (Musculoskeletal and connective tissue disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
ROTARY CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1
RESPIRATORY INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 1
CEREBRAL HAEMORRHAGE (Vascular disorders) | 1
CEREBRAL INFARCTION (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Viviant Tablet 20 mg (N=3423)
INSOMNIA (Psychiatric disorders) | 3
CRAMPS LEGS (Nervous system disorders) | 3
DIZZINESS (Nervous system disorders) | 5
DIZZINESS POSTURAL (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 6
SPINAL STENOSIS (Nervous system disorders) | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
PALPITATION (Cardiac disorders) | 5
EYE PAIN (Eye disorders) | 2
RETINAL HAEMORRHAGE (Eye disorders) | 1
VISION ABNORMAL (Eye disorders) | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 7
COLONIC POLYP (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 4
DIARRHOEA (Gastrointestinal disorders) | 4
DYSPEPSIA (Gastrointestinal disorders) | 51
ERUCTATION (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 3
MOUTH DRY (Gastrointestinal disorders) | 8
NAUSEA (Gastrointestinal disorders) | 13
VOMITING (Gastrointestinal disorders) | 3
ALLERGIC REACTION (General disorders) | 1
ASTHENIA (General disorders) | 1
CHEST DISCOMFORT (General disorders) | 2
EFFECT, LACK OF (General disorders) | 1
FACE OEDEMA (General disorders) | 2
FEVER (General disorders) | 2
LEG PAIN (General disorders) | 3
MALAISE (General disorders) | 1
OEDEMA (General disorders) | 2
OEDEMA GENERALISED (General disorders) | 2
OEDEMA PERIORBITAL (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 6
TEMPERATURE CHANGED SENSATION (General disorders) | 2
HEPATIC CYST (Hepatobiliary disorders) | 1
HEPATOCELLULAR DAMAGE (Hepatobiliary disorders) | 1
PHOSPHATASE ALKALINE INCREASED (Hepatobiliary disorders) | 2
SGOT INCREASED (Hepatobiliary disorders) | 1
SGPT INCREASED (Hepatobiliary disorders) | 1
BRONCHITIS (Infections and infestations) | 1
CYSTITIS (Infections and infestations) | 1
PHARYNGITIS (Infections and infestations) | 6
PNEUMONIA (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
LACERATION (Injury, poisoning and procedural complications) | 1
HYPERLIPAEMIA (Metabolism and nutrition disorders) | 1
OBESITY CENTRAL (Metabolism and nutrition disorders) | 1
WEIGHT INCREASE (Metabolism and nutrition disorders) | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
FRACTURE (Musculoskeletal and connective tissue disorders) | 2
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 6
DYSURIA (Renal and urinary disorders) | 1
RENAL CYST (Renal and urinary disorders) | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1
URINE ABNORMAL (Renal and urinary disorders) | 1
BREAST ENGORGEMENT (Reproductive system and breast disorders) | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 2
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
COUGHING (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
LARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
SPUTUM DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 8
RASH (Skin and subcutaneous tissue disorders) | 5
SKIN REACTION LOCALISED (Skin and subcutaneous tissue disorders) | 1
SWEATING INCREASED (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 5
FLUSHING (Vascular disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT01793142/Prot_SAP_000.pdf